CLINICAL TRIAL: NCT00108199
Title: Generalization of Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MHBS-001-01S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; vocational rehabilitation; neuropsychology
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Behavioral: Problem-Solving Training
Behavioral: Work-Related Social Skills Training

SUMMARY:
This study examines whether patients with schizophrenia can benefit from a problem-solving training intervention and whether a work-related social skills training intervention leads to improvements in the patient's performance at work.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with schizophrenia or schizoaffective disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States